CLINICAL TRIAL: NCT01495585
Title: Treatment of Chronic Delta Hepatitis With Lonafarnib
Brief Title: Lonafarnib for Chronic Hepatitis D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 120046; 12-DK-0046 (Other: NIH Clinical Center)
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Results first posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-07

CONDITIONS: Hepatitis D
Keywords: Hepatitis; Delta; Treatment; Lonafarnib; Hepatitis D
MeSH Terms: conditions — Hepatitis D; Hepatitis | interventions — lonafarnib

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo control
  Interventions: Other: Placebo
- Group 1 (Experimental): lonafarnib 100mg
  Interventions: Drug: Lonafarnib
- Group 2 (Experimental): lonafarnib 200mg
  Interventions: Drug: Lonafarnib

INTERVENTIONS:
Drug: Lonafarnib — Commercially approved products used to test the research hypothesis
  Arms: Group 1; Group 2
Other: Placebo — Placebo control
  Arms: Placebo

SUMMARY:
Background:

* Chronic hepatitis D is a severe disease of the liver caused by infection with the hepatitis D virus. The hepatitis D virus can only infect a person who also has hepatitis B; therefore, people with delta hepatitis have both hepatitis B and hepatitis D virus infection. Most people with hepatitis D eventually develop cirrhosis, which causes scarring and damage to the liver. There is currently no effective treatment for chronic hepatitis D.
* Lonafarnib is a drug that was originally designed to treat different types of cancer. It may be able to prevent the hepatitis D virus from reproducing itself. However, it has not been tested on people with hepatitis D. Researchers want to study different doses of lonafarnib to see how they affect virus levels and other symptoms of hepatitis D.

Objectives:

- To test the safety and effectiveness of lonafarnib as a treatment for chronic hepatitis D.

Eligibility:

- Individuals at least 18 years of age who have chronic hepatitis D.

Design:

* Participants will be screened with a medical history and physical exam. They will have blood and urine tests, eye exams, and imaging studies of the liver and gall bladder. A liver biopsy may also be performed.
* Participants will receive either lonafarnib or placebo twice a day for 28 days. For the first 3 days, participants will stay in the hospital to have frequent blood tests. Participants will have four more clinic visits (on days 7, 14, 21, and 28) for blood and urine tests. Eye exams and heart function tests will also be given. Men may be asked to provide sperm samples for further testing.
* After the 28 days of treatment, participants will stop taking the drug or placebo. They will have regular followup visits for up to 6 months after stopping treatment....

DETAILED DESCRIPTION:
Chronic delta hepatitis is a serious form of chronic liver disease caused by infection with the hepatitis D virus (HDV), a small RNA virus that requires farnesylation of its major structural protein (HDV antigen) for replication. We propose to treat between 12 and 14 patients with chronic delta hepatitis using the farnesyltransferase inhibitor (FTI) lonafarnib for a duration of twenty-eight days. Farnesyltransferase inhibitors have not been used in the therapy of delta hepatitis. Patients with HBsAg and HDV RNA in serum, elevated aminotransferases, or moderate-to-severe chronic hepatitis and HDV antigen on liver biopsy will be enrolled. Before receiving therapy, patients will be monitored for at least three months with regular testing for alanine aminotransferase (ALT) levels and will undergo Clinical Center admission for medical evaluation and percutaneous liver biopsy. Two dosing groups of lonafarnib will be assessed, with a placebo cohort in each group. At each clinic visit, patients will be questioned about side effects and symptoms, undergo focused physical examination, and have blood drawn for complete blood counts, HDV RNA, and routine liver tests (including ALT, AST, alkaline phosphatase, direct and total bilirubin, and albumin). At two-week intervals, for a period of 28 days, patients will also be tested for HBsAg, anti-HBs, HBV DNA, and prothrombin time. At the end of 28 days of treatment, patients will undergo repeat physical examination, assessment of symptoms (using a symptom scale questionnaire), complete blood counts, routine liver tests, and hepatitis B and D viral markers. The primary therapeutic endpoint will be an improvement in quantitative serum HDV RNA levels after 28 days of lonafarnib therapy. The primary safety endpoint will be the ability to tolerate the drug at the prescribed dose for the 4 week duration. Several secondary endpoints will be measured, including side effects, ALT levels, and symptoms. Therapy will be stopped for intolerance to lonafarnib (which will be carefully defined). This study is designed as a phase 2a study assessing the safety, tolerance and antiviral activity of two dose levels of lonafarnib, a farnesyltransferase inhibitor.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 18 years or above, male or female.
  2. Serum alanine or aspartate aminotransferase activities above the upper limit of normal (ALT > 41 or AST > 31 U/L) on an average of three determinations taken during the previous 6 months. The mean of the three determinations will be defined as baseline levels.
  3. Presence of anti-HDV in serum.
  4. Evidence of chronic hepatitis on liver biopsy done within the previous 12 months with a necroinflammatory score in histology activity index of at least 5 (out of a maximum of 18) and at least 1 for hepatic fibrosis (out of a maximum of 6).
  5. Presence of HDV antigen in liver tissue or HDV RNA in serum.
  6. Written informed consent.

EXCLUSION CRITERIA:

1. Decompensated liver disease, defined by bilirubin > 4mg/dL, albumin < 3.0 gm/dL, prothrombin time > 2 sec prolonged, or history of bleeding esophageal varices, ascites or hepatic encephalopathy. Laboratory abnormalities that are not thought to be due to liver disease may not necessarily require exclusion. Patients with ALT levels greater than 1000 U/L (> 25 times ULN) will not be enrolled but may be followed until three determinations are below this level.
2. Pregnancy or inability to practice adequate contraception, in women of childbearing potential or in spouses of such women. Adequate contraception is defined as vasectomy in men, tubal ligation in women, or use of two barrier methods such as condoms and spermicide combination, birth control pills, an intrauterine device, Depo-Provera, or Norplant.
3. Significant systemic or major illnesses other than liver disease, including, but not limited to, congestive heart failure, renal failure (eGFR < 50 ml/min), organ transplantation, serious psychiatric disease or depression (only if felt to be at high risk by the NIH psychiatric consultation service), and active coronary artery disease.
4. Systemic immunosuppressive therapy within the previous 2 months.
5. Evidence of another form of liver disease in addition to viral hepatitis (for example autoimmune liver disease, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson disease, alcoholic liver disease, nonalcoholic steatohepatitis (but not steatosis), hemochromatosis, or alpha-1-antitrypsin deficiency).
6. Active substance abuse, such as alcohol, inhaled or injection drugs within the previous year.
7. Evidence of hepatocellular carcinoma.
8. Evidence of concurrent hepatitis C infection with positive serum HCV RNA.
9. Any experimental therapy apart from pegylated interferon within 6 months prior to enrollment.
10. Diagnosis of malignancy in the five years prior to the enrollment with exception granted to superficial dermatologic malignancies.
11. Evidence of HIV co-infection; HIV (Omega) antibody positivity on serum testing.
12. Concurrent usage of statins as these drugs inhibit mevalonate synthesis which reduces protein prenylation.
13. Concurrent usage of moderate and strong CYP3A inhibitors and inducers.
14. Inability to understand or sign informed consent.
15. Any other condition, which in the opinion of the investigators would impede the patient s participation or compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theo Heller, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data with outside collaborators

REFERENCES:
- [Background] Glenn JS, Marsters JC Jr, Greenberg HB. Use of a prenylation inhibitor as a novel antiviral agent. J Virol. 1998 Nov;72(11):9303-6. doi: 10.1128/JVI.72.11.9303-9306.1998. PMID 9765479
- [Background] Rizzetto M, Ponzetto A, Forzani I. Hepatitis delta virus as a global health problem. Vaccine. 1990 Mar;8 Suppl:S10-4; discussion S21-3. doi: 10.1016/0264-410x(90)90207-3. PMID 2183511
- [Background] Rosina F, Rizzetto M. Treatment of chronic type D (delta) hepatitis with alpha interferon. Semin Liver Dis. 1989 Nov;9(4):264-6. doi: 10.1055/s-2008-1040521. No abstract available. PMID 2690350
- [Derived] Kefalakes H, Koh C, Sidney J, Amanakis G, Sette A, Heller T, Rehermann B. Hepatitis D Virus-Specific CD8+ T Cells Have a Memory-Like Phenotype Associated With Viral Immune Escape in Patients With Chronic Hepatitis D Virus Infection. Gastroenterology. 2019 May;156(6):1805-1819.e9. doi: 10.1053/j.gastro.2019.01.035. Epub 2019 Jan 18. PMID 30664876
- [Derived] Koh C, Canini L, Dahari H, Zhao X, Uprichard SL, Haynes-Williams V, Winters MA, Subramanya G, Cooper SL, Pinto P, Wolff EF, Bishop R, Ai Thanda Han M, Cotler SJ, Kleiner DE, Keskin O, Idilman R, Yurdaydin C, Glenn JS, Heller T. Oral prenylation inhibition with lonafarnib in chronic hepatitis D infection: a proof-of-concept randomised, double-blind, placebo-controlled phase 2A trial. Lancet Infect Dis. 2015 Oct;15(10):1167-1174. doi: 10.1016/S1473-3099(15)00074-2. Epub 2015 Jul 16. PMID 26189433
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-DK-0046.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Group 1, participants were randomized either placebo or lonafarnib 100 mg. In Group2, participants were randomized into either placebo or lonafarnib 200 mg.
Groups:
- Placebo: Two placebo participants in Group1 and two placebo participants in Group 2. The two placebo participants in Group 1 received open label lonafarnib 200 mg.
- Lonafarnib 100 mg: 6 participants were randomized to Lonafarnib 100 mg.
- Lonafarnib 200 mg: 4 participants were randomized to Lonafarnib 200 mg.
Period: Overall Study
Arm/Group | Placebo | Lonafarnib 100 mg | Lonafarnib 200 mg
Started | 4 | 6 | 4
Open Label Lonafarnib 200 mg | 2 | 0 | 0
Completed | 4 | 6 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled patients were sequentially assigned into one of two dosing groups which consisted of lonafarnib 100mg in group 1 and lonafarnib 200mg in group 2, with placebo controls in each group.
  Group1 placebo patients received open-label lonafarnib as group 2 participants.
Groups:
- Lonafarnib 200 mg: 4 participants were randomized to Lonafarnib 200 mg and two "Placebo" participants in Lonafarnib 100 mg arm received open label lonafarnib 200 mg .
- Total: Total of all reporting groups
Arm/Group | Placebo | Lonafarnib 100 mg | Lonafarnib 200 mg | Total
Number analyzed (Participants) | 4 | 6 | 6 | 16
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [33 to 39] | 36 [30 to 42] | 45 [38 to 55] | 38 [33 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 5
  Male | 2 | 5 | 4 | 11
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 26.5 [24.1 to 28.9] | 22.8 [21.9 to 23.5] | 26.1 [25.5 to 27.3] | 24.4 [21.9 to 27.3]
Pre-treatment mucleoside analogues [Number; unit: participants]
  yes | 1 | 2 | 2 | 5
  no | 3 | 4 | 4 | 11
Ethnic origin [Number; unit: participants]
  Asian | 2 | 3 | 3 | 8
  White | 1 | 3 | 3 | 7
  African | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Quantitative Serum HDV RNA Levels After 28 Days of Lonafarnib Therapy.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: log(IU/ml)
Groups:
- Placebo: placebo control.
  Group 1 placebo participants received open-label lonafarnib as group 2 participants.
  Each group consisted of 8 participants (6 lonafarnib ands 2 placebo).
- Group 1: lonafarnib 100 mg
- Group 2: lonafarnib 200 mg
Arm/Group | Placebo | Group 1 | Group 2
Number analyzed (Participants) | 4 | 6 | 6
log(IU/ml) | -0.13 (0.14) | -0.73 (0.54) | -1.54 (0.36)
Statistical Analysis 1: Comparison: Placebo vs Group 1; Student t-test was used on the change in serum log HDV RNA after 28 days of therapy with lonafarnib; Test type: Superiority or Other; p = 0.03, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Group 2; Student t-test was used on the change in serum log HDV RNA after 28 days of therapy with lonafarnib; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: ALT Levels
Time Frame: 7 months
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Group 1 | Group 2
Number analyzed (Participants) | 4 | 6 | 6
U/L | 18 (13) | 4 (93) | 29 (85)
Statistical Analysis 1: Comparison: Placebo vs Group 1; Test type: Superiority or Other; p = 0.96, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Group 2; Test type: Superiority or Other; p = 0.6, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Placebo | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/4 | 6/6 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | Group 1 (N=6) | Group 2 (N=6)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 6 (6)
Decreased appetite (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (5)
Abdominal bloating/dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 6 (6)
Vomitting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Weight loss > 2kg (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 6 (6)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (General disorders) | 1 (1) | 1 (1) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Lightheadedness (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes